CLINICAL TRIAL: NCT00551720
Title: Motivation and Patch Treatment for HIV-positive Smokers
Acronym: Positive PATHS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA012344 (NIH)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections; Smoking Cessation
Keywords: HIV; HIV positive; AIDS; smoking cessation; smoking; smoking counseling
MeSH Terms: conditions — HIV Infections; Smoking Cessation; HIV Seropositivity; Acquired Immunodeficiency Syndrome; Smoking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (Experimental)
  Interventions: Behavioral: Standard Care
- Motivational Enhancement (Experimental)
  Interventions: Behavioral: Motivational Enhancement

INTERVENTIONS:
Behavioral: Standard Care — Brief advice and follow-up provided a smoking-cessation trained Health Educator PLUS nicotine patch
  Arms: Standard Care
Behavioral: Motivational Enhancement — Brief advice and follow-up, nicotine patch, and the addition of a tailored motivational intervention and behavioral skills counseling for smoking cessation.
  Arms: Motivational Enhancement

SUMMARY:
The purpose of this study is to develop and evaluate a brief, clinic-based smoking cessation treatment for an HIV+ population. We compared two treatments, a brief advice and follow-up plus nicotine patch treatment(Standard Care; SC) and brief advice and follow-up, nicotine patch, with the addition of a tailored motivational intervention and behavioral skills counseling for smoking cessation (Motivationally-Enhanced; ME), in a randomized controlled trial. We hypothesized that those HIV+ participants receiving the ME will demonstrate greater biochemically verified smoking abstinence rates at 6-month follow-up than those receiving the SC control treatment. All study participants were offered use of the nicotine patch.

DETAILED DESCRIPTION:
Cigarette smoking is highly prevalent among HIV+ individuals, posing unique health risks, impacting HAART-therapy effectiveness, and possibly altering the course of the disease. To our knowledge, Motivation and Patch Treatment for HIV-Positive Individuals (Positive PATHS) was the first NIH-funded smoking cessation intervention designed to motivate HIV+ smokers to quit. Participants were referred by physicians at eight Immunology clinics in New England and randomized to receive either a brief, two-session intervention (Standard Care; SC) modeled on PHS guidelines, or a more intensive, four-session motivational counseling intervention (Motivational-Enhancement; ME). All physicians participating in the trial were trained in study eligibility criteria, as well as basic smoking cessation counseling strategies (based on the PHS guidelines). Interested individuals were then referred to the study, with a study researcher explaining the details of the study and obtaining informed consent. Participants were then assisted in completing baseline assessments via laptop computer, and then randomized to receive either a brief intervention (2-sessions) designed to reflect the standard of care in outpatient hospital settings and modeled on PHS guidelines (standard care; SC) or a more intensive (4-session) motivational counseling intervention (motivational enhancement; ME), with both interventions providing 8-weeks of nicotine replacement (patches; NRT) to those participants willing to set a quit date. Follow-up assessments, including biochemical verification of self-reported quitters (via carbon monoxide measurement) were conducted at 2, 4, and 6 months from baseline. This study is among the first to examine the health effects of a delivered smoking cessation intervention to an HIV+ population, with the results having implications for treatments in clinical care settings.

ELIGIBILITY:
Inclusion Criteria:

* Be receiving care for HIV at one of the participating immunology clinics
* Be 18 years old or older
* Be current (past 7 days) cigarette smoker
* Speak English or Spanish

Exclusion Criteria:

* Are pregnant or nursing
* Have uncontrolled hypertension
* Use other forms of tobacco like cigars or chewing tobacco or are using anything else to help with quitting smoking
* Are allergic to the nicotine patch or have a skin condition like eczema or psoriasis that makes them unable to use the patch

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 1999-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
smoking cessation | 6-months

SECONDARY OUTCOMES:
smoking cessation | 2- and 4-months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Niaura, PhD, Principal Investigator — Brown University-Butler Hospital; Elizabeth Lloyd-Richardson, PhD, Study Director — Brown University/The Miriam Hospital
Locations (5):
- United States (5):
  - Stanley Street Treatment and Resources, Inc., Fall River, Massachusetts
  - Greater New Bedford Community Center, New Bedford, Massachusetts
  - Hope Center for HIV Care, Memorial Hospital, Pawtucket, Rhode Island
  - Rhode Island Hospital HIV Clinic, Providence, Rhode Island
  - The Miriam Hospital Immunology Clinic, Providence, Rhode Island

REFERENCES:
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] Lloyd-Richardson EE, Stanton CA, Papandonatos GD, Shadel WG, Stein M, Tashima K, Flanigan T, Morrow K, Neighbors C, Niaura R. Motivation and patch treatment for HIV+ smokers: a randomized controlled trial. Addiction. 2009 Nov;104(11):1891-900. doi: 10.1111/j.1360-0443.2009.02623.x. Epub 2009 Aug 28. PMID 19719796